CLINICAL TRIAL: NCT07088484
Title: Watch-and-Wait Strategy in Patients With Objective Response After Immuno-chemotherapy for Locally Recurrent Nasopharyngeal Carcinoma: A Prospective Multicenter Observational Study
Brief Title: Watch-and-Wait After Immunochemotherapy in Locally Recurrent Nasopharyngeal Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: lrNPCimmuno
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
Keywords: locally recurrent nasopharyngeal carcinoma, watch-and-wait strategy, immuno-chemotherapy, low-intensity maintenance treatment
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICI-chemotherapy cohort: All included patients will undergo protocolized ICI-chemotherapy for 4-6 cycles, following by LIMT.
  Interventions: Drug: ICI-chemotherapy and LIMT

INTERVENTIONS:
Drug: ICI-chemotherapy and LIMT — gemcitabine, docetaxel, paclitaxel, cisplatin, platinum, capecitabine, S1; Tislelizumab.

SUMMARY:
The purpose of this study is to compare chemotherapy plus immunotherapy with immunochemotherapy combined subsequent locoregional radiotherapy in recurrent nasopharyngeal carcinoma (NPC), in order to confirm the value of immunotherapy and chemotherapy in recurrent NPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, regardless of sex.
2. Treatment-naïve patients with newly diagnosed metastatic nasopharyngeal carcinoma (NPC).
3. Receiving immunotherapy. (or Treated with immunotherapy)
4. At least one measurable tumor lesion according to RECIST (Response Evaluation Criteria in Solid Tumors) version 1.1.
5. Adequate organ function.
6. Signed and dated informed consent form indicating that the patient (or legally authorized representative) has been informed of all pertinent aspects of the study.
7. Patients willing and able to comply with scheduled visits and study procedures.

Exclusion Criteria:

1. Patients with distant metastasis of nasopharyngeal carcinoma.
2. Patients who have not received immunotherapy or chemotherapy. (Alternatively: No prior immunotherapy or chemotherapy.)
3. History of another active malignancy within the past 5 years, except for malignancies with a negligible risk of metastasis or death (e.g., expected 5-year overall survival >90%) or malignancies treated with curative intent and with no evidence of disease (e.g., adequately treated carcinoma in situ of the cervix, basal cell or squamous cell carcinoma of the skin, localized prostate cancer treated with curative intent, ductal carcinoma in situ of the breast treated surgically with curative intent).
4. Lack of capacity to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All included patients will undergo protocolized ICI-chemotherapy for 4-6 cycles, following by LIMT, with the local treatment be postponed or omitted.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | Counting from the start of the treatment for two years.
  Defined as the time from the initiation of ICI-chemotherapy to disease progression or death for any reason, whichever occurred first.

IPD SHARING:
Plan to Share IPD: Undecided